CLINICAL TRIAL: NCT04805242
Title: Effects of Dextrose Prolotherapy in Rotator Cuff Disease: A Randomized Controlled Study
Brief Title: Effects of Dextrose Prolotherapy in Rotator Cuff Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Selim Sezikli, MD, Principal Investigator, Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Shoulder Prolotherapy
Record Dates: First submitted 2021-03-12; First posted 2021-03-18 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Rotator Cuff Disease
Keywords: Rotator Cuff Disease; Dextrose Prolotherapy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dextrose prolotherapy groups (Active Comparator): In the first group, dextrose prolotherapy injection will be applied.
  Interventions: Other: Dextrose Prolotherapy Injection
- Saline groups (Sham Comparator): In the second group, physiological saline injection will be applied.
  Interventions: Other: Saline Injection

INTERVENTIONS:
Other: Dextrose Prolotherapy Injection — Subacromial injection: 5 cc solution (15% dextrose + saline + 1% lidocaine solution) will be injected into the subacromial bursa using a sterile 21 gauge injector.
  Extra-articular injection: Previously marked using a sterile 27 gauge injector (dental needle); A total of 10 cc solution (15% dextrose + saline + 1% lidocaine solution) will be injected into the infraspinatus, teres minor, supraspinatus insertion on the tuberculum majus, the subscapularis insertion on the tuberculum minus, the coracoid process and the long head of the biceps.
  As a home exercise program, shoulder range of motion and stretching, shoulder isometric and isotonic strengthening exercises will be given at least three days a week with 3 sets of 10 repetitions.
  Arms: Dextrose prolotherapy groups
Other: Saline Injection — Subacromial injection: 5 cc solution (saline + 1% lidocaine solution) will be injected into the subacromial bursa using a sterile 21 gauge injector.
  Extra-articular injection: 5 cc solution (saline + 1% lidocaine solution) will be injected to the attachment areas of the previously marked tendons to the bone using a sterile 30 gauge injector.
  As a home exercise program, shoulder range of motion and stretching, shoulder isometric and isotonic strengthening exercises will be given at least three days a week with 3 sets of 10 repetitions.
  Arms: Saline groups

SUMMARY:
The aim of this prospective, randomized, controlled, single-blind study is to determine the effects of dextrose prolotherapy on shoulder pain and functions in patients with chronic rotator cuff disease.

DETAILED DESCRIPTION:
Rotator cuff disease is a major cause of shoulder pain and disability. Non-surgical treatments to reduce pain and improve function have included therapeutic exercises, NSAIDs, subacromial corticosteroid injections. However, some patients are resistant to these conservative treatments. In recent years, prolotherapy has increased in popularity for the treatment of musculosketal conditions. Regenerative injection methods can be applied in resistant chronic rotator cuff disease. In this prospective, randomized controlled, single blind, interventional study, a total of 60 patients with shoulder pain due to rotator cuff disease who meet eligibility criteria will be enrolled in the study. Eligible participants will be randomly assigned to one of the two groups using computer-generated random numbers. In the dextrose prolotherapy group, ultrasound-guided prolotherapy injections will be applied under aseptic conditions at 0, 3, and 6 weeks. In the salin injection group, salin injections will be applied under aseptic conditions at 0, 3, and 6 weeks. Home exercise program will be apply to both groups. Participants are going to evaluate before injection, and at the 1-month follow-up and 3-month follow-up using the visual analog scale (VAS) scores for pain during activity, at rest, and at night, with the Shoulder Pain and Disability Index (SPADI) change in pain and disability score, with The University of California and Los Angeles Rating Score (UCLA) change in pain and functional score and the change in the Ultrasound Shoulder Pathology Rating Scale (USPRS).

ELIGIBILITY:
Inclusion Criteria:

* Shoulder pain for more than 3 months
* Being resistant to conservative treatment for at least 3 months
* Being in the age range of 30-65
* Presence of rotator cuff disease detected in current magnetic resonance imaging and confirmed by clinical examination.

Exclusion Criteria:

* Presence of rheumatic disease or other systemic inflammatory diseases
* Having a diagnosis of uncontrolled diabetes mellitus
* Evidence of infection (systemically or locally on the shoulder)
* The presence of a previous operation on the shoulder
* Bleeding tendency (acquired or hereditary) [INR> 2 in the patient using coumadin]
* Injected shoulder within the previous 8 weeks
* The presence of local anesthesia and corn allergy
* Passive shoulder abduction <100 ° or external rotation <25 °
* Rotator cuff calcification diameter> 0.8cm in current direct graph or Usg
* Presence of serious comorbidity

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-11-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline activity pain score at 1-months and 3-months | Baseline, 1-month, 3-month
  Visual Analogue Scale-Activity pain (0-10 point). Higher scores mean a worse outcome

SECONDARY OUTCOMES:
Change from baseline rest pain score at 1-months and 3-months | Baseline, 1-month, 3-month
  Visual Analogue Scale-Rest pain (0-10 point). Higher scores mean a worse outcome
Change from baseline night pain score at 1-months and 3-months | Baseline, 1-month, 3-month
  Visual Analogue Scale-Night pain (0-10 point). Higher scores mean a worse outcome
Change from baseline pain, disability at 1-months and 3-months | Baseline, 1-month, 3-month
  Shoulder Pain and Disability Index (SPADI) measures shoulder pain and disability. It consists of 2 chapters and 13 subtitles in total. The total score range in the scale varies between 0-130. High scores are associated with more pain, and disability, while low scores indicate well-being.
Change from baseline shoulder pain and function at 1-months and 3-months | Baseline, 1-month, 3-month
  UCLA Shoulder Rating Score (The University of California and Los Angeles Rating Score); Over a total of 35 points, pain, function, patient satisfaction, flexion muscle strength, flexion angle are evaluated. Pain and function are evaluated on a scale of 1-10 points each, active flexion angle, flexion muscle strength, and patient satisfaction on a scale of 1-5 points each. In total, 34-35 points are considered excellent, 29-33 points good, and values below 29 points are considered poor. This outcome measure is a composite outcome measure consisting of multiple measures.
Change from baseline rotator cuff structure at 1-months and 3-months | Baseline, 1-month, 3-month
  USPRS (Ultrasound Shoulder Pathology Rating Scale); It is a scale that enables the evaluation of rotator cuff structures using ultrasound. It is evaluated over 20 points. High scores indicate increased pathology severity.
Change from baseline shoulder flexion muscle strenght and flexion angle at 1-months and 3-months | Baseline, 1-month, 3-month
  UCLA Shoulder Rating Score (The University of California and Los Angeles Rating Score); Over a total of 35 points, pain, function, patient satisfaction, flexion muscle strength, flexion angle are evaluated. Pain and function are evaluated on a scale of 1-10 points each, active flexion angle, flexion muscle strength, and patient satisfaction on a scale of 1-5 points each. In total, 34-35 points are considered excellent, 29-33 points good, and values below 29 points are considered poor.
Change from baseline patient satisfaction at 1-months and 3-months | Baseline, 1-month, 3-month
  UCLA Shoulder Rating Score (The University of California and Los Angeles Rating Score); Over a total of 35 points, pain, function, patient satisfaction, flexion muscle strength, flexion angle are evaluated. Pain and function are evaluated on a scale of 1-10 points each, active flexion angle, flexion muscle strength, and patient satisfaction on a scale of 1-5 points each. In total, 34-35 points are considered excellent, 29-33 points good, and values below 29 points are considered poor.
Change from baseline shoulder range of motion at 1-months and 3-months | Baseline, 1-month, 3-month
  Shoulder range of motion was measured using a goniometer

CONTACTS AND LOCATIONS:
Overall Officials: Selim Sezikli, MD, Principal Investigator — Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation; Demirhan Diracoglu, Prof., Study Director — Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation
Locations (1):
- Istanbul University Istanbul Faculty of Medicine, Department of Physical Medicine and Rehabilitation, Istanbul, Fatih, Turkey (Türkiye)